CLINICAL TRIAL: NCT06011252
Title: Pacing Characteristics of a Conventional Bipolar, Active Fixation Pacing Lead for Left Bundle Branch Area Pacing in Patients With Symptomatic Bradycardia
Brief Title: Pacing Characteristics of a Conventional Bipolar
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200877A3
Record Dates: First submitted 2023-07-28; First posted 2023-08-25 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Symptomatic Bradycardia
Keywords: FF068; Conventional bipolar; symptomatic bradycardia; left bundle branch area pacing; LBBAP

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, multi-center, non-randomized, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Solia S lead with any BIOTRONIK Pacemaker (Other): * Name: Solia S lead with any BIOTRONIK Pacemaker
  * Model: Solia S45/S53/S60
  * Manufacturer: BIOTRONIK SE & Co. KG
  * Method of use: LBBAP implantation for all bradycardia indications.
  * Mechanism of action: (1) Pacemaker stimulates the cardiac tissue to keep stable heart beats in patients with bradycardia. (2) LBBAP can be an alternative to right ventricular (RV) pacing to reduce RV pacing-induced ventricular dyssynchrony.
  * Device category and grade: E3610 Cardiovascular devices, Class III
  Interventions: Device: Solia S lead with any BIOTRONIK Pacemaker

INTERVENTIONS:
Device: Solia S lead with any BIOTRONIK Pacemaker — * Name: Solia S lead with any BIOTRONIK Pacemaker
  * Model: Solia S45/S53/S60
  * Manufacturer: BIOTRONIK SE & Co. KG
  * Method of use: LBBAP implantation for all bradycardia indications.
  * Mechanism of action: (1) Pacemaker stimulates the cardiac tissue to keep stable heart beats in patients with bradycardia. (2) LBBAP can be an alternative to right ventricular (RV) pacing to reduce RV pacing-induced ventricular dyssynchrony.
  * Device category and grade: E3610 Cardiovascular devices, Class III

SUMMARY:
Study Title:

Pacing characteristics of a conventional bipolar, active fixation pacing lead for left bundle branch area pacing in patients with symptomatic bradycardia

Study Objectives:

To characterize an approach for left bundle branch area pacing (LBBAP) in patients with bradycardia indications for pacing and to assess implant success rate, safety, and long-term stability with a conventional bipolar, active fixation pacing lead.

Methodology: Open-label, prospective, multi-center, non-randomized, single-arm study

Study Endpoints:

Primary Endpoint:

• Implant success rate

Secondary Endpoints:

* Intra-operative procedure time and fluoroscopic exposure time
* Intra-operative intracardiac electrogram (EGM) changes: paced QRS duration, stimulus to left ventricular (LV) activation time, and LBB potential
* Post-operative imaging data: posteroanterior, left anterior oblique 30O, right anterior oblique 30O, Left lateral views
* Serial paced 12-lead electrocardiogram (ECG) and intracardiac EGM changes: QRS duration (QRSd), pacing-QRS interval, and new atrial ﬁbrillation (AF)
* Serial echocardiography changes: left ventricular ejection fraction (LVEF), left atrial (LA) and LV chamber size, and global longitudinal strain (GLS) of tissue Doppler imaging
* Serial changes of pacing parameters: capture threshold, impedance, and sensing amplitude for both atrial and ventricular Solia S leads
* Safety:

Immediate (< 24 hours), in-hospital, and chronic (12 months) adverse events

DETAILED DESCRIPTION:
Patient Enrollment: To target 120 consecutive patients while considering a 20% dropout rate, an approximate sample size of 150 patients is needed.

Treatment Plan:This is a prospective, single-arm, open-label, non-randomized, multi-center study to investigate the feasibility and stability of left bundle branch area pacing (LBBAP) for ventricular pacing in symptomatic bradycardia patients with a conventional bipolar, active fixation pacing lead. Eligible patients will be enrolled through the process of informed consent in the seven clinical investigational sites across Taiwan with competitive enrollment.

All subjects enrolled in the study will undergo LBBAP implantation using one or two Solia S leads in combination with any legally marketed BIOTRONIK pacemaker system delivered through a preshaped sheath (Selectra 3D) via left cephalic, left subclavian, or left axillary venous access. The available lengths of Solia S are 45, 53, and 60 cm. As for which one will be used, it will depend on the lead configuration and the anatomy of the subject. During the screening period, the subject's medical history and demographic information will be collected. The baseline data will be obtained prior to the pacing implantation. Depending on the needs of the subject, the screening and implantation procedures may be performed on the same day. Implant data will include lead measurements, implant technique, and lead positioning. After completion of pacemaker implantation, subjects will be followed at 1, 3, 6, and 12 months or until lead failure (dislodgment, high capture threshold, or inadequate sensing requiring revision of the lead) or death. During follow-up, a determination will be made whether the system is able to provide appropriate pacing and sensing.

Device Description:

Solia Leads: The Solia S is a family of 5.6 French, steroid-eluting, transvenous, endocardial, bipolar active fixation leads with an extendable/retractable and electrically active screw. The Solia S is manufactured, like its predecessor, the Siello S lead, in three different models (45, 53, and 60 cm in length). It has an isodiametric structure and silicone insulation. The inner and outer conductors consist of quadruple wire coils.

Solia S has a diameter of 5.6 F and is covered by a polyurethane overlay for improved gliding. It has an IS-1 connector and a 10 mm pole distance. The area between tip and ring is flexible in order to minimize the perforation risk. The fixation screw of the Solia S is electrically active and has a fractal iridium coating. The screw can be extended by 1.8 mm and has an active surface area of 4.5 mm2. The ring electrode of Solia S has a surface area of approximately 17.4 mm2 and is fractally coated with iridium. The Solia S has a dexamethasone eluting steroid collar containing 0.85 mg dexamethasone acetate. The accessories that are delivered with the lead are identical to the accessories of the Siello S.

Test Device information is below,

* Name: Solia S lead with any BIOTRONIK Pacemaker
* Model: Solia S45/S53/S60
* Manufacturer: BIOTRONIK SE & Co. KG
* Method of use: LBBAP implantation for all bradycardia indications.
* Mechanism of action: (1) Pacemaker stimulates the cardiac tissue to keep stable heart beats in patients with bradycardia. (2) LBBAP can be an alternative to right ventricular (RV) pacing to reduce RV pacing-induced ventricular dyssynchrony.
* Device category and grade: E3610 Cardiovascular devices, Class III

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 20 years of age
* Standard bradycardia pacing indications requiring new ventricular lead implantation
* Able to give informed consent for the participation in the trial

Exclusion Criteria:

* Patients underwent cardiac resynchronization therapy or implantable cardioverter-defibrillator implantation
* New York Heart Association (NYHA) functional class IV heart failure
* Life expectancy < 1 year
* Right-sided approach for lead implantation
* Hemodialysis or peritoneal dialysis patients
* Pregnant or breast-feeding women
* Abnormal baseline findings considered by the investigator to indicate conditions that might affect study endpoints
* Participation in another prospective interventional clinical study within a period of 4 weeks prior to the implantation of LBBAP
* Use of any recreational drugs or history of drug addiction
* Any other condition that, in the investigator's judgment, might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Implant Success Rate | Baseline, 12 months
  The purpose of the primary endpoint is to evaluate the overall success rate of the implanted system, including Solia ventricular lead to sense and deliver pacing at 12- month post-implant. Successful sensing performance at 12 months is the demonstrated ability to appropriately sense without intervention for undersensing (i.e., Solia leadrelated adverse event for lead undersensing or loss of sensing) in the period from implant to 12 months, except for normal pulse generator reprogramming. Successful pacing is the demonstrated ability at 12 months to deliver a stimulation pulse with capture, without intervention (i.e., Solia lead-related adverse event for intermittent capture or no lead capture) other than normal pulse generator reprogramming. Success is determined at the subject level.

SECONDARY OUTCOMES:
Intra-operative fluoroscopic exposure time | Baseline, 1 months, 3 months, 6 months ,and 12 months
  Fluoroscopic exposure time will be measured and recorded during the LBBAP implantation period.
Intra-operative intracardiac electrogram (EGM) | Baseline, 1 months, 3 months, 6 months ,and 12 months
  Intra-operative intracardiac electrogram will be measured and recorded at baseline & during LBBAP implantation. Paced QRS duration, stimulus to left ventricular (LV) activation time, and LBB potential will be recorded if feasible.
  The data are included: Heart Rate (bpm) & QRSd (ms) & PR interval (ms) & QTc interval (ms)
Post-operative imaging data | baseline
  X-Ray imaging data is included posteroanterior view, left anterior oblique (30 degree) view, right anterior oblique (30 degree) view, Left lateral views will be collected after LBBAP implantation.
Serial paced 12-lead electrocardiogram (ECG) and intracardiac EGM changes | Screen, Baseline, 1 months, 3 months, 6 months ,and 12 months
  During implantation and follow-up periods, a 12-lead ECG will be recorded along with an intracardiac EGM. The QRS duration (QRSd), pacing-QRS interval, and imaging data, new atrial fibrillation on the surface ECG will be collected and analyzed.
  ECG will be recorded with paced AV interval 100ms or sensed AV interval 60ms in patients with intact AV conduction if possible.
Serial echocardiography changes | baseline, 12 months
  Echocardiography will be performed at baseline and 12-months postimplant to evaluate the changes of the left ventricular ejection fraction (LVEF), left atrial (LA), and left ventricular (LV) chamber size, tissue Doppler global longitudinal strain (GLS) from baseline. Thedata are including LVEF (%) & LVEDD (mm) & LAD (mm) & LVESD (mm) & IVS (mm) & LVPW (mm)
Serial changes of pacing parameters | Baseline, 1 months, 3 months, 6 months ,and 12 months
  Pacing parameters, including capture threshold, impedance, and sensing amplitude for both atrial and ventricular Solia S leads will be collected and evaluated at baseline, 1-month, 3-month, 6-month, and 12-months post-implant. Capture threshold measurement will be performed at 0.4 ms pulse width when feasible. The data are including Basic Rate: (min) & Rest Rate: (min) & Max Rate: (min) Paced AV delay (ms) & Sensed AV delay (ms) & Atrial lead: sensitivity (mV); output _ V@_____ ms & Ventricular lead: sensitivity (mV) ; output ______ V@_____ ms

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chieh Wang, Principal Investigator — Chang Gung Memorial Hospital
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital, Linkou District, Taipei
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - MacKay Memorial Hospital, Taipei
  - National Yang Ming Chiao Tung University Hospital, Yilan